CLINICAL TRIAL: NCT03188042
Title: A Multi-site Interventional Pilot Study Using Transorbital Alternating Current Stimulation for People With Glaucoma
Brief Title: A Study Using Transorbital Alternating Current Stimulation for People With Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-02005
Record Dates: First submitted 2017-06-01; First posted 2017-06-15 (Actual); Results first posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Glaucoma
Keywords: Transorbital Alternating Current Stimulation; Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- rtACS Stimulation Group (Experimental)
  Interventions: Device: rtACS Stimulation
- Sham Intervention Group (Sham Comparator): Sham stimulation looks like rtACS, but is not active rtACS.
  Interventions: Device: Sham Intervention

INTERVENTIONS:
Device: rtACS Stimulation — Electric current stimulation; rtACS is a non-invasive application of electric current to stimulate the retina to induce synaptic efficacy, in particular those cells that have some measure of dysfunction but are not dead, and oscillations of nearby neuronal ensembles.
  Arms: rtACS Stimulation Group
Device: Sham Intervention — A computer-controlled sham stimulation function for masking interventionist to study group. The device will be used to deliver a weak electric current stimulation protocol to participants via electrodes placed transorbitally, with one reference electrode positioned elsewhere.
  Arms: Sham Intervention Group

SUMMARY:
This pilot study will test the preliminary efficacy and feasibility of an intervention protocol for one method of electric current stimulation, repetitive transorbital alternating current stimulation (rtACS), to treat visual impairment in people with glaucoma. We will evaluate a study protocol to use in future clinical trials to test the effectiveness of rtACS to ameliorate the progressive effects of vision loss both structurally and functionally in the eye, the visual pathway, and in regard to people's independence (i.e., functional ability). In this prospective, randomized controlled, double-masked pilot study, we will: 1) determine an effect of rtACS on ophthalmic structure and function (from retina to visual brain), 2) assess the methodology of procedures for assessment of people's functional ability and quality of life (QoL) to determine an effect of rtACS, and 3) assess the feasibility and implementation of the pilot study protocol for a larger multi-site, randomized controlled trial.

DETAILED DESCRIPTION:
Participants will engage in baseline, intervention, post-intervention, and follow-up visits over the span of approximately 8 weeks. The expected outcomes for this project are that (1) rtACS activates viable but poorly or non-functional retinal ganglion cells to improve their structural and functional capabilities, (2) measures of retinal, optic nerve, and visual brain structures and function will correspond with improvement in visual function, and (3) changes in visual function following rtACS will be associated with improvements in participants' functional ability and QoL. rtACS has successfully been used in the rehabilitation of visual impairments in people with optic neuropathies; however, we do not know the clinical value of rtACS specifically for people with glaucoma, including the effect of rtACS on people's functional ability and QoL.

ELIGIBILITY:
Inclusion Criteria:

* Live in a community, residential setting (i.e., non-institutionalized, not homeless)
* Diagnosis of glaucoma (not type-specific, excluding traumatic glaucoma): Moderate defect or worse in both eyes but not total blindness
* Visual field defects present for at least 6 months
* Best-corrected visual acuity of 20/200 (1.0 logMAR) or better in at least one eye
* Commitment to comply with study procedures (2 week period of intervention sessions) with baseline, post-intervention, and follow-up visits

Exclusion Criteria:

* Other optic comorbidity than glaucoma
* End-stage organ disease or medical condition with subsequent vision loss (e.g., diabetes, stroke)
* Other diseases of the retina or cataracts responsible for worse than 20/70 best-corrected visual acuity
* Photosensitivity to flickering lights
* Intraocular Pressure (IOP) > 27 mmHg at baseline

  * Medically diagnosed memory disorder or Telephone Interview for Cognitive Status-modified (TICS-m) score ≤ 27
* Electric or electronic implants (e.g., cardiac pacemaker)
* Metallic artifacts/implants in head and/or torso
* Diagnosed epilepsy
* Epileptic seizure within the past 3 years of enrollment date
* Auto-immune disease, acute stage (e.g., rheumatoid arthritis)
* Metastatic disease
* Certain mental diseases/psychiatric conditions (e.g., schizophrenia) that would preclude reliable testing and participation
* Unstable medical conditions (e.g., diabetes, diabetes causing diabetic retinopathy)
* Claustrophobia (to limit functional neuroimaging)
* Received rtACS in the past

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Schuman, MD, FACS, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Ramos Cadena MLA, Sohn A, Livengood H, Lee TF, Rubin B, Hu J, Sabel BA, Matayev R, Panarelli J, Wollstein G, Schuman JS. Transorbital Alternating Current Stimulation in a Double-Masked Randomized Clinical Trial: Visual Functional Effect and Quality of Life. Ophthalmol Sci. 2024 Sep 4;5(1):100614. doi: 10.1016/j.xops.2024.100614. eCollection 2025 Jan-Feb. PMID 39584183

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Started | 8; 16 Eyes | 10; 20 Eyes
Completed | 7; 14 Eyes | 9; 18 Eyes
Not Completed | 1; 2 Eyes | 1; 2 Eyes
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rtACS Stimulation Group | Sham Intervention Group | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10) | 59 (20) | 61 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 9 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Peripapillary RNFL Thickness
Description: Peripapillary retinal nerve fiber layer (RNFL) thickness (μm) measured using optical coherence tomography (OCT).
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: micrometers (μm)
Units Other Than Participants: Eyes
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 7 | 9
Number analyzed (Eyes) | 14 | 18
micrometers (μm) | -0.13 (2.3) | -1.8 (3.91)

2. Primary Outcome: Change in Macular Ganglion Cell-Inner Plexiform Layer Thickness
Description: Macular ganglion cell-inner plexiform layer thickness (μm) measured using OCT.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: micrometers (μm)
Units Other Than Participants: Eyes
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 7 | 9
Number analyzed (Eyes) | 14 | 18
micrometers (μm) | -0.13 (0.99) | 0.3 (4.52)

3. Primary Outcome: Percentage Change in ON Head Cup-to-Disc Ratio
Description: Percentage change in optic nerve (ON) head cup-to-disc ratio measured using OCT.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: percentage (%) change
Units Other Than Participants: Eyes
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 7 | 9
Number analyzed (Eyes) | 14 | 18
percentage (%) change | 0 (0.01) | 0.01 (0.01)

4. Primary Outcome: Change in Humphrey Visual Field Analyzer Score
Description: The Humphrey Visual Field Analyzer assesses the mean deviation (dB), a measure of visual field sensitivity through threshold testing. dBs tested by the Humphrey analyzer range between 0 and 50 dB (0 is the brightest and 50 is the dimmest). A value of 0 means the patient could not see the brightest target, and a 50 means the dimmest target was seen. Most values are around 30 dB, and any numbers below this range imply a possible visual field defect.
Time Frame: Baseline, Week 4
Measure: Median (Standard Deviation); unit: dB
Units Other Than Participants: Eyes
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 7 | 9
Number analyzed (Eyes) | 14 | 18
dB | 0.86 (6.27) | 2.89 (9.65)

5. Primary Outcome: Change in Score on Assessment of Life Habits (LIFE-H), Short Form 3.1
Description: The LIFE-H short form 3.1 is a 77-item questionnaire developed to measure: (1) how a respondent accomplishes regular activities and social roles and (2) respondent's satisfaction with how regular activities and social roles are accomplished. The LIFE-H total score is obtained by summing the scores on each item and then dividing by the number of items. The LIFE-H score ranges from 0 to 9, where a score of 0 indicates total handicap or total disruption in participation and a score of 9 means an optimal level of participation.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 7 | 9
score on a scale | 0.000137 (0.165273) | -0.089842 (0.150235)

6. Primary Outcome: Change in Minnesota Low Vision Reading Test (MNRead): Reading Acuity Score
Description: An estimate of reading acuity is given by the smallest print size at which the patient can read the entire sentence without making significant errors. This method measures acuity to the nearest 0.1 logMAR. Each sentence in the MNRead Reading Acuity chart has 60 characters, which corresponds to 10 standard length words, assuming a standard word length of 6 characters (including a space). Reading acuity is calculated as follows: Reading acuity = size of smallest sentence read + 0.01 x number of errors.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 7 | 9
Number analyzed (Eyes) | 14 | 18
logMAR | -0.02857 (0.108233) | 0.013333 (0.074498)

7. Primary Outcome: Change in Score on National Eye Institute Visual Functioning Questionnaire (VFQ-39)
Description: National Eye Institute VFQ-39 measures health-related quality of life in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, peripheral vision, and composite score. For each domain: the lowest and highest possible scores are 0 and 100 points, respectively. Higher score means higher functioning. The total score is the average of the domain scores.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 7 | 9
score on a scale | 3.52 (2.1405453) | 0.95 (0.089)

8. Primary Outcome: Change in Score on 36-Item Short Form Survey (SF-36)
Description: The SF-36 is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state. The total score is the average of the domain scores.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 7 | 9
score on a scale | 23.14 (5.3030631) | 17.18 (0.1888264)

9. Primary Outcome: VEP-Measured Amplitude (15% Contrast) at Baseline
Description: Visual evoked potential (VEP) identifies decreased visual function and helps with discriminations of glaucomatous changes by measuring amplitude (micro volts) and latency (milliseconds (ms)) with 15% contrast parameters.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: micro volts
Units Other Than Participants: Eyes
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 3 | 4
Number analyzed (Eyes) | 6 | 8
micro volts | 5.675 (3.208632886) | 10.6655 (2.1296074)

10. Primary Outcome: VEP-Measured Latency (15% Contrast) at Baseline
Description: as for outcome 9
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Units Other Than Participants: Eyes
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 3 | 4
Number analyzed (Eyes) | 6 | 8
milliseconds | 119.166667 (26.759733) | 130.75 (19.70828929)

11. Primary Outcome: VEP-Measured Amplitude (85% Contrast) at Baseline
Description: Visual evoked potential (VEP) identifies decreased visual function and helps with discriminations of glaucomatous changes by measuring amplitude (micro volts) and latency (milliseconds (ms)) with 85% contrast parameters.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: micro volts
Units Other Than Participants: Eyes
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 5 | 6
Number analyzed (Eyes) | 10 | 12
micro volts | 8.3314 (2.794988157) | 10.0365 (3.7914384)

12. Primary Outcome: VEP-Measured Latency (85% Contrast) at Baseline
Description: as for outcome 11
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Units Other Than Participants: Eyes
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 5 | 6
Number analyzed (Eyes) | 10 | 12
milliseconds | 110.5 (11.051018) | 121 (10.839742)

13. Primary Outcome: VEP-Measured Amplitude (15% Contrast) at Week 4
Description: as for outcome 9
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: micro volts
Units Other Than Participants: Eyes
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 4 | 5
Number analyzed (Eyes) | 8 | 10
micro volts | 6.62025 (0.905566995) | 7.1814 (2.865013)

14. Primary Outcome: VEP-Measured Latency (15% Contrast) at Week 4
Description: as for outcome 9
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: milliseconds
Units Other Than Participants: Eyes
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 4 | 5
Number analyzed (Eyes) | 8 | 10
milliseconds | 119.25 (11.97566978) | 131.7 (14.267971)

15. Primary Outcome: VEP-Measured Amplitude (85% Contrast) at Week 4
Description: as for outcome 11
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: micro volts
Units Other Than Participants: Eyes
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 6 | 5
Number analyzed (Eyes) | 12 | 10
micro volts | 8.4108333 (4.3606635) | 9.8224 (2.8729446)

16. Primary Outcome: VEP-Measured Latency (85% Contrast) at Week 4
Description: as for outcome 11
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: milliseconds
Units Other Than Participants: Eyes
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 6 | 5
Number analyzed (Eyes) | 12 | 10
milliseconds | 119.4166667 (11.8634593) | 122.3 (10.556988)

17. Primary Outcome: Pelli-Robson Contrast Sensitivity Chart Score at Baseline
Description: The Pelli-Robson test measures contrast sensitivity using a single large letter size (20/60 optotype), with contrast varying across groups of letters. The chart uses letters (6 per line), arranged in groups whose contrast varies from high to low. Patients read the letters, starting with the highest contrast, until they are unable to read two or three letters in a single group. A score is assigned based on the contrast of the last group in which two or three letters were correctly read. The score, a single number, is a measure of the subject's log contrast sensitivity. A Pelli-Robson score of 2.0 indicates normal contrast sensitivity of 100 percent. Scores less than 2.0 signify poorer contrast sensitivity. Pelli-Robson contrast sensitivity score of less than 1.5 is consistent with visual impairment and a score of less than 1.0 represents in visual disability.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: LogCS
Units Other Than Participants: Eyes
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 7 | 9
Number analyzed (Eyes) | 14 | 18
LogCS | 1.4 (0.42) | 1.26 (0.47)

18. Primary Outcome: Pelli-Robson Contrast Sensitivity Chart Score at Week 4
Description: as for outcome 17
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: LogCS
Units Other Than Participants: Eyes
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 7 | 9
Number analyzed (Eyes) | 14 | 18
LogCS | 1.39 (0.35) | 1.08 (0.55)

19. Primary Outcome: Early Treatment Diabetic Retinopathy Study (ETDRS) Visual Acuity Score (VAS) at Baseline
Description: ETDRS charts have five Sloan letters on each line; the lines are of equal difficulty, and there is a geometric progression in letter size from line to line. Beginning with Chart 1, the right eye is tested with the left eye occluded. Following the completion of testing the right eye, the left eye is tested with Chart 2 while covering the right eye. Each letter is scored as right or wrong. Correct letters are circled on the scoresheet. Each letter read correctly is assigned a score and each line is totaled at the end of testing. VAS awards one point for every letter correctly guessed. The total scores range from 0 to 100, with higher scores indicating greater visual acuity.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 7 | 9
Number analyzed (Eyes) | 14 | 18
score on a scale | 0.08 (0.13) | 0.16 (0.16)

20. Primary Outcome: Early Treatment Diabetic Retinopathy Study (ETDRS) Visual Acuity Score (VAS) at Week 4
Description: as for outcome 19
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
Number analyzed (Participants) | 7 | 9
Number analyzed (Eyes) | 14 | 18
score on a scale | 0.10 (0.14) | 0.16 (0.17)

ADVERSE EVENTS:
Description: Adverse event data were not collected from participants in this study.
Arm/Group | rtACS Stimulation Group | Sham Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT03188042/Prot_SAP_000.pdf